CLINICAL TRIAL: NCT03644238
Title: The Acute Effect of Physical Activity on Blood Glucose in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: OGTT study
Record Dates: First submitted 2018-04-09; First posted 2018-08-23 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Glucose Tolerance Test; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental intervention (Experimental): Oral Glucose Tolerance Test and physical activity
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test; Behavioral: Physical activity
- Control intervention (Other): Oral Glucose Tolerance Test and inactivity.
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test; Behavioral: Inactivity

INTERVENTIONS:
Diagnostic Test: Oral Glucose Tolerance Test — 75g of glucose is consumed
  Other Names: OGTT
Behavioral: Inactivity — Lying or sitting down.
  Arms: Control intervention
Behavioral: Physical activity — 20 minutes of fixed intensity exercise on a bicycle ergometer.
  Arms: Experimental intervention

SUMMARY:
The aim of the project is to investigate the acute effect of exercise on blood glucose after glucose consumption. Thereby we wish to achieve knowledge that can improve prevention and treatment of gestational overweight and gestational diabetes mellitus (GDM). This will prevent serious complications during pregnancy and birth, but also long term complications like type 2 diabetes mellitus (T2DM) for both the mother and the offspring.

15 pregnant participants will perform two Oral Glucose Tolerance Tests (OGTT). One is followed by physical activity and the other is followed by inactivity and will serve as control. Blood glucose will be monitored continuously during the study.

DETAILED DESCRIPTION:
Cases: 15 pregnant women recruited at the routine ultrasound scan at gestational week 19 at the Department of Obstetrics and Gynecology, Aarhus University Hospital. Subjects will receive both written and oral information before entering the trial. Subjects with a prepregnancy BMI > 27 and no other risk factors of diabetes will be included in the study. The women will be examined during gestational week 27-30 where the routine Oral Glucose Tolerance Test (OGTT) will take place. The routine OGTT will serve as control.

Intervention: The subjects will perform two OGTT separated by a minimum of two days. One - the regular OGTT will serve as control and the second OGTT will be the intervention. The two days in between will function as a "wash out period" to avoid potential carry over effect. During the OGTT subjects will consume a liquid containing 75g of glucose. The control OGTT will be followed by inactivity. The intervention OGTT will be immediately followed by 20 minutes of exercise on a bicycle ergometer with a fixed intensity.

Study variables: Blood glucose will be monitored continuously using the IPro2 Continous Glucose Monitor (CGM) from Medtronic. A sensor is inserted into interstitial fluid and continuously generates an electrical current proportional to the glucose concentration. A recorder stores the average sensor current every 5 minutes.

In both control and intervention, blood tests will be taken at time 0, 1 and 2 hours after the OGTT. Blood samples will be analyzed for blood glucose, HbA1c, C-peptide and insulin.

Data on demography, family history of diabetes, prepregnancy BMI, gestational weight gain and complications during pregnancy are collected from medical records of the patients and their offspring.

ELIGIBILITY:
Inclusion Criteria:

* Prepregnancy BMI > 27

Exclusion Criteria:

* Physical disability that affect movement

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Blood glucose | Through intervention periods of 2 hours.
  Difference in blood glucose between experimental intervention and control intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Per Ovesen, MD, Prof., Study Director — Aarhus University Hospital / University of Aarhus
Locations (1):
- Department of Obstetrics and Gynecology, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andersen MB, Ovesen PG, Daugaard M, Ostenfeld EB, Fuglsang J. Cycling reduces blood glucose excursions after an oral glucose tolerance test in pregnant women: a randomized crossover trial. Appl Physiol Nutr Metab. 2020 Nov;45(11):1247-1252. doi: 10.1139/apnm-2020-0020. Epub 2020 May 22. PMID 32442384